CLINICAL TRIAL: NCT00017212
Title: A Phase II Study Of Intravenous Exatecan Mesylate (DX-891F) Administered Daily For Five Days Every Three Weeks To Patients With Previously Untreated Metastatic Gastric Cancer
Brief Title: DX-8951f in Treating Patients With Metastatic Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068663; DAIICHI-8951A-PRT028; SACI-IDD-00-27; UTHSC-0015011134
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of exatecan mesylate in treating patients who have metastatic stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate of patients with previously untreated metastatic gastric cancer treated with exatecan mesylate (DX-8951f).
* Determine the time to tumor progression in this patient population when treated with this drug.
* Determine the survival at 6 and 12 months in this patient population when treated with this drug.
* Determine the quantitative and qualitative toxic effects of this drug in this patient population.
* Determine the pharmacokinetics of this drug in the plasma of these patients.

OUTLINE: This is a multicenter study.

Patients receive exatecan mesylate (DX-8951f) IV over 30 minutes on days 1-5. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric or gastroesophageal adenocarcinoma

  * Lymph node involvement and/or distant metastasis
* No squamous cell carcinoma, small cell carcinoma, lymphoma, or leiomyosarcoma of the stomach
* Measurable disease with indicator lesions outside the field of prior radiotherapy

  * At least 20 mm by conventional scan OR
  * At least 10 mm by spiral CT scan
  * Nonmeasurable lesions include the following:

    * Primary tumor
    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonitis
    * Cystic lesions
    * Abdominal masses not confirmed and followed by imaging techniques
* No prior treatment for locally advanced or metastatic disease

  * Prior adjuvant treatment allowed if disease recurrence noted at least 6 months after completion of adjuvant treatment
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST or ALT no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* Albumin at least 2.8 g/dL
* PT or INR no greater than 1.5 times ULN (coumadin independent)

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction within the past 6 months

Other:

* No concurrent serious infection
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No overt psychosis, mental disability, or incompetence that would preclude informed consent
* No other life-threatening illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Biologic therapy:

* No concurrent anti-cancer biologic therapy
* No concurrent prophylactic colony stimulating factors during first course of therapy

Chemotherapy:

* Recovered from prior adjuvant chemotherapy
* No other concurrent anti-cancer chemotherapy
* No other concurrent anti-cancer cytotoxic therapy

Endocrine therapy:

* Concurrent megestrol for appetite stimulation allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy and recovered
* No prior wide-field radiotherapy to more than 25% of bone marrow
* No concurrent anti-cancer radiotherapy

Surgery:

* At least 4 weeks since prior major surgery and recovered
* No concurrent anti-cancer surgery

Other:

* No other investigational drugs (including analgesics or antiemetics) for at least 4 weeks prior to, during, and for 4 weeks after study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (6):
- United States (5):
  - Pacific Shores Medical Group, Long Beach, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
- Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Ajani JA, Takimoto C, Becerra CR, Silva A, Baez L, Cohn A, Major P, Kamida M, Feit K, De Jager R. A phase II clinical and pharmacokinetic study of intravenous exatecan mesylate (DX-8951f) in patients with untreated metastatic gastric cancer. Invest New Drugs. 2005 Oct;23(5):479-84. doi: 10.1007/s10637-005-2907-z. PMID 16133799